CLINICAL TRIAL: NCT02924064
Title: Efficacy and Safety of Teneligliptin in Combination With Metformin in Chinese Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MP-513-C03
Record Dates: First submitted 2016-09-26; First posted 2016-10-05 (Estimated); Results first posted 2022-01-28 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — 3-(4-(4-(3-methyl-1-phenyl-1H-pyrazol-5-yl)piperazin-1-yl)pyrrolidin-2-ylcarbonyl)thiazolidine; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Teneligliptin 20mg (Experimental): Teneligliptin (20mg once daily) for 24 weeks in combination with metformin
  Interventions: Drug: Teneligliptin 20mg; Drug: Metformin ≥ 1000 mg
- Placebo (Placebo Comparator): Placebo for 24 weeks in combination with metformin
  Interventions: Drug: Placebo; Drug: Metformin ≥ 1000 mg

INTERVENTIONS:
Drug: Teneligliptin 20mg
  Arms: Teneligliptin 20mg
Drug: Placebo
  Arms: Placebo
Drug: Metformin ≥ 1000 mg

SUMMARY:
This study is designed as a prospective, multi-centre, parallel group, double-blind randomized, placebo-controlled, phase 3 clinical study to evaluate the efficacy and safety of MP-513 (Teneligliptin) in combination with metformin.

ELIGIBILITY:
Inclusion Criteria:

* A signed and dated informed consent form obtained from the subject, in accordance.
* The subject is aged ≥18 years at signature of the informed consent form.
* Hospitalization status: outpatient.
* The subject has a documented diagnosis of type 2 diabetes mellitus for at least 3 months at the screening visit (Day -28).
* The subject's type 2 diabetes mellitus is managed by metformin monotherapy ≥1000 mg/day plus diet and exercise therapy, and the dosage or dose regimen of metformin and diet and exercise regimen has not been changed for at least 8 consecutive weeks at the screening visit (Day -28). Subjects who cannot do exercise due to complication are not limited to this criteria.
* The subject's HbA1c is ≥ 7.0% and < 10.0% at the screening visit (Day -28) and on Day -14.

Exclusion Criteria:

* The subject has a history of type 1 diabetes mellitus or a secondary form of diabetes.
* The subject has received insulin within 1 year prior to the screening visit (Day -28), with the exception of insulin therapy during hospitalization or insulin therapy for medical conditions not requiring hospitalization (< 2 weeks' duration).
* The subject has received an anti-diabetic drug within 8 weeks prior to the screening visit (Day -28).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2016-09; Primary Completion 2018-09-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: General Manager, Study Director — Tanabe Pharma Corporation
Locations (1):
- Investigational center, Beijing, China

RESULTS

PARTICIPANT FLOW:
Groups:
- Teneligliptin 20mg + Metformin: Teneligliptin (20 mg once daily) for 24 weeks in combination with metformin.
- Placebo + Metformin: Placebo for 24 weeks in combination with metformin.
Period: Overall Study
Arm/Group | Teneligliptin 20mg + Metformin | Placebo + Metformin
Started | 123 | 124
FAS | 122 | 124
Completed | 99 | 81
Not Completed | 24 | 43
Not completed — Adverse Event | 2 | 2
Not completed — Lost to Follow-up | 0 | 2
Not completed — Physician Decision | 0 | 2
Not completed — Protocol Violation | 1 | 3
Not completed — Withdrawal by Subject | 4 | 5
Not completed — Other | 17 | 29

BASELINE CHARACTERISTICS:
Population: FAS: All subjects in the randomized set who have received at least one dose of study medication during the double-blind treatment period and have at least one post-baseline efficacy observation. Subjects who were not diagnosed with type 2 diabetes mellitus were excluded.
Groups:
- Total: Total of all reporting groups
Arm/Group | Teneligliptin 20mg + Metformin | Placebo + Metformin | Total
Number analyzed (Participants) | 122 | 124 | 246
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.0 (9.8) | 54.7 (10.1) | 55.3 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 57 | 98
  Male | 81 | 67 | 148
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 122 | 124 | 246
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Changes in HbA1c at Week 24
Description: The change in HbA1c from baseline to Week 24 in Teneligliptin compared to Placebo was performed on FAS.
Time Frame: at Day 1(baseline) and Week 24
Population: All subjects in the randomized set who have received at least one dose of study medication during the double-blind treatment period and have at least one post-baseline efficacy observation. Subjects who were not diagnosed with type 2 diabetes mellitus were excluded.
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | Teneligliptin 20mg + Metformin | Placebo + Metformin
Number analyzed (Participants) | 122 | 124
percentage of HbA1c | -0.72 (0.07) | -0.01 (0.07)

2. Secondary Outcome: The Changes in Fasting Plasma Glucose (FPG) at Week 24
Description: The change in FPG from baseline to Week 24 in Teneligliptin compared to Placebo was performed on FAS.
Time Frame: at Day 1(baseline) and Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Teneligliptin 20mg + Metformin | Placebo + Metformin
Number analyzed (Participants) | 122 | 124
mg/dL | -13.5 (3.3) | 3.0 (3.3)

ADVERSE EVENTS:
Time Frame: 24 weeks
Description: All subjects in the randomized set who have received at least one dose of study medication during the double-blind treatment period. One subject who had been randomized in placebo group was handled as Teneligliptin group, because the subject had been administered Teneligliptin mistakenly.
Arm/Group | Teneligliptin 20mg + Metformin | Placebo + Metformin
All-Cause Mortality (participants affected / at risk) | 0/124 | 0/123
Serious Adverse Events (participants affected / at risk) | 4/124 | 6/123
Other Adverse Events (participants affected / at risk) | 35/124 | 43/123
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Teneligliptin 20mg + Metformin (N=124) | Placebo + Metformin (N=123)
Arrhythmia (Cardiac disorders) | 0 | 1
Sinus node dysfunction (Cardiac disorders) | 0 | 1
Cataract (Eye disorders) | 0 | 1
Gastric polyps (Gastrointestinal disorders) | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 2 | 1
Hypertension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Teneligliptin 20mg + Metformin (N=124) | Placebo + Metformin (N=123)
Upper respiratory tract infection (Infections and infestations) | 14 | 22
Hyperlipidaemia (Metabolism and nutrition disorders) | 8 | 7
Hyperuricaemia (Metabolism and nutrition disorders) | 11 | 13
Proteinuria (Renal and urinary disorders) | 7 | 5
Hypertension (Vascular disorders) | 3 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2016-04-29): https://cdn.clinicaltrials.gov/large-docs/64/NCT02924064/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-11): https://cdn.clinicaltrials.gov/large-docs/64/NCT02924064/SAP_001.pdf